CLINICAL TRIAL: NCT05742269
Title: Molecular PD-L1 PET/CT Imaging With 89Zr-atezolizumab to Monitor Immune Responses in Metastatic Triple Negative Breast Cancer
Brief Title: Molecular PD-L1 PET/CT Imaging With 89Zr-atezolizumab in Metastatic Triple Negative Breast Cancer
Acronym: MIMIR-mTNBC
Status: Recruiting | Type: Observational
Sponsor: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Renske Altena, Principal Investigator, Karolinska University Hospital
Other Study IDs: MIMIR-mTNBC
Record Dates: First submitted 2023-01-17; First posted 2023-02-23 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Metastatic Triple-Negative Breast Carcinoma
Keywords: 89Zr-atezolizumab; PD-L1 PET; predictive biomarker
MeSH Terms: conditions — Triple Negative Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- PD-L1 positive disease (on PET and/or IHC): Nab-paclitaxel at a dose of 100 mg per square meter of body-surface area, administered intravenously, on days 1, 8, and 15, and carboplatin at a dose of Area Under the Curve (AUC) 5 on day 1 of every 28-day cycle.
  The patients with a PD-L1+ tumour, according to IHC with the SP142 antibody (≥ 1% on immune cells) and/or 89Zr-atezolizumab tracer uptake on PET-imaging, will receive atezolizumab at a dose of 840 mg, administered intravenously, on days 1 and 15.
  Interventions: Diagnostic Test: 89Zr-atezolizumab PET/CT
- PD-L1 negative disease (on PET and IHC): Nab-paclitaxel at a dose of 100 mg per square meter of body-surface area, administered intravenously, on days 1, 8, and 15, and carboplatin at a dose of Area Under the Curve (AUC) 5 on day 1 of every 28-day cycle.
  Interventions: Diagnostic Test: 89Zr-atezolizumab PET/CT

INTERVENTIONS:
Diagnostic Test: 89Zr-atezolizumab PET/CT — All patients undergo a 89Zr-atezolizumab PET/CT. Allocation to chemotherapy + atezolizumab in case of a PD-L1 positive tumor (on IHC and/or PET)

SUMMARY:
The overarching purpose of this study is to improve precision medicine through more refined therapy selection for breast cancer patients who are candidates for ICI therapy (monoclonal antibodies targeting the programmed death ligand 1 (PD-L1) or programmed cell death protein 1 (PD-1)). The reference standard biomarker for ICI therapy selection is PD-L1 protein expression measured by immunohistochemistry (IHC). Several disadvantages exist with this method, the most important ones being inter- and intralesional as well as spatial heterogeneity in PD-L1 expression, as well as the need for invasive procedures to obtain material for analysis. The study hypothesis is that Positron Emission Tomography combined with Computed Tomography (PET/CT) imaging with a contemporary radiotracer (89Zr-atezolizumab), visualizing PD-L1 expression in the whole body, could be a better predictive biomarker to select which patients benefit from ICI. The use of PET/CT imaging with new radiotracers enables a non-invasive assessment of the presence of the target of treatment in the whole body and provides the possibility to combine functional information with anatomical details.

DETAILED DESCRIPTION:
Patients with mTNBC scheduled for first line palliative systemic treatment with nab-paclitaxel and carboplatin can be included. This chemotherapy combination is used to maximize the therapeutic potential of this first line systemic treatment line, extrapolating signals from early TNBC and in the absence of signs that indicate augmented safety issues.

The investigational medical product is 89Zr-atezolizumab. The pharmaceutical preparation of the IMP consists of the precursor atezolizumab combined with zirconium-89 to form 89Zr-atezolizumab. The radiolabelling of atezolizumab will be performed at the Department of Radiopharmacy, Karolinska University Hospital, Solna. This involves an automated synthesis procedure in a Good Manufacturing Practice facility.

All patients are scheduled for treatment with nab-paclitaxel at a dose of 100 mg per square meter of body-surface area, administered intravenously, on days 1, 8, and 15, and carboplatin at a dose of Area Under the Curve (AUC) 5 on day 1 of every 28-day cycle. The patients with a PD-L1+ tumour according to IHC with the SP142 antibody (≥ 1% on immune cells) and/or 89Zr-atezolizumab tracer uptake on PET-imaging, will receive atezolizumab at a dose of 840 mg, administered intravenously, on days 1 and 15.

ELIGIBILITY:
Inclusion Criteria:

* Patients with metastatic triple negative breast cancer (mTNBC), defined by pathological criteria: oestrogen receptor expression <10%, progesterone receptor expression <10%, HER2 negative, on the primary tumour or a metastatic biopsy
* Measurable disease according to RECIST v1.1
* At least one metastatic lesion accessible for biopsy
* Deemed by treating physician as fit for systemic therapy according to study protocol
* ECOG performance score 0/1
* Age ≥ 18 years old
* Adequate blood tests for bone marrow, renal and hepatic functions
* Able and willing to provide written informed consent

Exclusion Criteria:

* Previous treatment with chemotherapy or targeted therapy for mTNBC. Radiation therapy and previous chemotherapy (including taxanes) in the context of curative therapy is allowed.
* Contraindications for PET/CT as defined for clinical practice
* Other malignancy diagnosed within the last five years, except for radically treated basal or squamous cell carcinoma of the skin or CIS of the cervix
* Patients in child-bearing age without adequate contraception. Examples of contraceptive methods with a failure rate of < 1% per year include bilateral tubal ligation, male sterilization, established, proper use of hormonal contraceptives that inhibit ovulation, hormone-releasing intrauterine devices (IUDs), and copper IUDs. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not acceptable methods of contraception. Women must refrain from donating eggs during this same period.
* Pregnancy or lactation
* Uncontrolled hypertension, heart-, liver-, or kidney-diseases or other medical/psychiatric disorders.
* History of autoimmune disease, including but not limited to myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjögren's syndrome, Guillain-Barré syndrome, multiple sclerosis, vasculitis, or glomerulonephritis

  * Patients with a history of autoimmune-related hypothyroidism on a stable dose of thyroid replacement hormone are eligible for this study. Patients with controlled Type 1 diabetes mellitus on a stable insulin regimen may be eligible for this study.
  * Patients with eczema, psoriasis, lichen simplex chronicus or vitiligo with dermatologic manifestations only (e.g., no psoriatic arthritis) are permitted provided that they meet the following conditions: Rash must cover less than 10% of body surface area (BSA); Disease is well controlled at baseline and only requiring low potency topical steroids; No acute exacerbations of underlying condition within the last 12 months (not requiring PUVA [psoralen plus ultraviolet A radiation], methotrexate, retinoids, biologic agents, oral calcineurin inhibitors, high potency or oral steroids).
* Vaccination with a live vaccine within 30 days of the first dose of study treatment
* A known history of Human Immunodeficiency Virus (HIV) infection, hepatitis B (HBsAg reactive) or hepatitis C (HCV RNA detected) infection or active tuberculosis.
* Treatment with systemic corticosteroids or other systemic immunosuppressive medications (including but not limited to prednisone, dexamethasone, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor [TNF] agents) within 2 weeks prior to randomization, or anticipated requirement for systemic immunosuppressive medications during the trial

  * Patients who have received acute, low-dose, systemic immunosuppressant medications (e.g., a one-time dose of dexamethasone for nausea) may be enrolled in the study
  * Patients with a history of allergic reaction to IV contrast requiring steroid pre-treatment should have baseline and subsequent tumor assessments performed using CT.
  * The use of inhaled corticosteroids for chronic obstructive pulmonary disease, mineralocorticoids (e.g., fludrocortisone) for patients with orthostatic hypotension, and low-dose supplemental corticosteroids for adrenocortical insufficiency are allowed.
* Hypersensitivity to atezolizumab

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with newly diagnosed irresectable or metastatic triple negative breast cancer
Sampling Method: Probability Sample
Enrollment: 64 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Level of statistical agreement (Cohen kappa coefficient) between PD-L1 status on IHC (with SP142 Ventana) and PET (with 89Zr-atezolizumab) | baseline
  Level of statistical agreement by means of Cohen's kappa coefficient between PD-L1 IHC (positive defined as expression ≥1% on immune cells with SP142) and PD-L1 PET/CT (PD-L1 positivity is defined as having at least one lesion with radiotracer uptake over the background uptake).
  Level of statistical agreement by means of Cohen's kappa coefficient between PD-L1 IHC (positive defined as expression ≥1% on immune cells with SP142) and PD-L1 PET/CT (PD-L1 positivity is defined as having at least one lesion with radiotracer uptake over the background uptake).
  Level of statistical agreement by means of Cohen's kappa coefficient between PD-L1 IHC (positive defined as expression ≥1% on immune cells with SP142) and PD-L1 PET/CT (PD-L1 positivity is defined as having at least one lesion with radiotracer uptake over the background uptake).

SECONDARY OUTCOMES:
Treatment outcomes - response rate | Baseline - up to one year
  Disease response rates in three patient groups
  1. IHC positive and PET positive,
  2. IHC positive and PET negative,
  3. IHC negative and PET positive.
Treatment outcomes - progression free survival | Baseline - up to one year
  Progression free survival in three patient groups
  1. IHC positive and PET positive,
  2. IHC positive and PET negative,
  3. IHC negative and PET positive.
Treatment-related toxicities | Baseline - up to one year
  Treatment discontinuation rates in three patient groups
  1. IHC positive and PET positive,
  2. IHC positive and PET negative,
  3. IHC negative and PET positive.
Heterogeneity in PD-L1 status | Baseline
  Discordance in 89Zr-atezolizumab between different sites and within metastatic sites in the body.
Improved staging | Baseline
  Percentage of 89Zr-atezolizumab uptake in sites, not previously determined on the routine radiological investigation with CT, as a measure of cancer spread determined on whole body 89Zr-atezolizumab PET/CT in and different metastases.

OTHER OUTCOMES:
Immune infiltrate and PD-L1 status | Baseline
  Differences in number of immune cells cells in biopsied sites with discordance between PD-L1 IHC and PD-L1 PET.
ICI toxicity prediction | Baseline - up to one year
  Rates (and severity according to CTC-AE) of immune-mediated side effects in relation to 89Zr-atezolizumab tracer uptake in organs at risk for immune-mediated toxicities.

CONTACTS AND LOCATIONS:
Overall Officials: Renske Altena, MD PhD, Principal Investigator — Karolinska Institutet; Jonas Bergh, MD, Prof, Study Director — Karolinska Institutet
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Undecided